CLINICAL TRIAL: NCT05917925
Title: Randomized, Double-blind Clinical Study to Evaluate the Effect of a Food Supplement Based on Hydrolyzed Collagen on Joint Function in a Moderately Active Population.
Brief Title: Evaluation of the Effect of a Food Supplement Based on Hydrolyzed Collagen on Joint Function.
Acronym: COLART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Francisco Javier Martínez Noguera (Other)
Collaborators: San Antonio Technologies - San Antonio Catholic University of Murcia (Other)
Responsible Party: Sponsor-Investigator, Francisco Javier Martínez Noguera, PhD (Head of the nutrition area of the Research Center for High Performance Sport), Universidad Católica San Antonio de Murcia
Organization: Universidad Católica San Antonio de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE012308
Record Dates: First submitted 2023-05-08; First posted 2023-06-26 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Pain, Acute; Pain, Chronic; Knee Osteoarthritis; Knee Injuries
Keywords: Hydrolyzed collagen; Post-exercise pain; Supplementation; Inflammation; Quality of life
MeSH Terms: conditions — Acute Pain; Chronic Pain; Osteoarthritis, Knee; Knee Injuries; Inflammation | interventions — Collagen

STUDY DESIGN:
Intervention Model Description: A randomized parallel study will be conducted in which 80 subjects will be divided into 2 groups: COL) 10 g/d hydrolyzed collagen-based supplement; PLA) 10 g/d placebo (maltodextrin) for 12 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COLLAGEN (COL) (Experimental): Subjects in this group will intake 10 g/day of a hydrolyzed collagen-based supplement.
  Interventions: Dietary Supplement: COLLAGEN (COL)
- PLACEBO (PLA) (Placebo Comparator): Subjects in this group will intake 10 g/day of placebo (maltodextrin).
  Interventions: Dietary Supplement: PLACEBO (PLA)

INTERVENTIONS:
Dietary Supplement: COLLAGEN (COL) — The collagen-based supplement will be ingested every day for 12 weeks at the same time.
  Arms: COLLAGEN (COL)
Dietary Supplement: PLACEBO (PLA) — The placebo will be ingested every day for 12 weeks at the same time.
  Arms: PLACEBO (PLA)

SUMMARY:
This clinical study evaluates the effect of taking a hydrolyzed collagen-based supplement on pain, function and quality of life in a moderately physically active population. Non-pathological knee pain is a common occurrence in many healthy people and can limit the quality of life. Therefore, the resolution of this problem can bring many benefits in terms of quality of life.

DETAILED DESCRIPTION:
Study design

Randomized, double-blind, placebo-controlled clinical trial with 2 parallel study groups (collagen-based formulation and placebo). Participants will take the study products for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who exercise regularly and meet the WHO definition of being moderately active.
* Persistent exercise-associated knee pain lasting at least 2 months prior to study inclusion.
* Knee pain score on the visual analogue pain scale of at least 30 mm, taking into account that the scale has a maximum range of 100 mm.

Exclusion Criteria:

* Individuals with severe illness.
* Subjects who are taking or have been treated within the last 7 days with glucosamine, chondroitin sulphate, collagen or hyaluronic acid injections or any dietary supplement indicated for joint health.
* Subjects with chronic inflammatory diseases affecting the musculoskeletal apparatus.
* Subjects with obesity (BMI ≥ 30 Kg/m2).
* Allergy or known hypersensitivity to any of the ingredients in the investigational product.
* Phenylketonuria.
* Treatment with narcotics, steroidal anti-inflammatory drugs or immunosuppressants. - Symptoms of extreme pain requiring high doses of analgesic therapy for a period of time longer than 2 weeks or intra-articular injection treatment.
* Individuals with diabetes.
* Pregnant women.
* Lactating women.
* Subjects who are participating in a clinical trial.
* Subjects who have participated in a clinical trial for pain in the last month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Intensity of knee pain | Throughout study completion, an average of 12 weeks
  It will be measured using a 100 mm long horizontal visual analogue scale (VAS) on which the participant must mark the pain he/she feels with 0 being "none" and 100 being "the most intense pain he/she can imagine". Once the level of pain is marked on the horizontal line, the length is measured from 0 in millimetres with a millimetre ruler.
  The results will be evaluated according to three levels of pain based on the marked values:
  <40 mm: Values below 40 mm indicate mild or mild moderate pain
  40-60 mm: If the measurement is between 40 and 60 mm, the pain is considered moderate to moderate-severe
  >60 mm: If the values are greater than 60 mm, the pain is considered severe to unbearable.

SECONDARY OUTCOMES:
Physical activity data | The following data will be recorded during the baseline visit
  Intensity by applying the IPAQ questionnaire and type (running, cycling, climbing, tennis, football...).
Demographic data | The following data will be recorded during the baseline visit
  Age, sex, employment status (active, unemployed, retired, student ....).
Frequency of alcohol and tobacco consumption | The following data will be recorded during the baseline visit
  Alcohol consumption and tobacco consumption (grams of alcohol and cigarettes per week)
Weight | The following data will be recorded during the baseline visit
  It will be measured by means of a precision balance (kg)
Height | The following data will be recorded during the baseline visit
  It will be measured by means of a stadiometer (cm)
Body mass index | The following data will be recorded during the baseline visit
  It will be calculated by the following formula kg/m2
Clinical data | The following data will be recorded during the baseline visit
  Symptoms are unilateral (Yes/No), Other joint problems (back, hand, neck, feet, shoulder, hip)
Current analgesic medication: | The following data will be recorded during the baseline visit
  Medication that has been taken at least once a week during the previous month. The name or active ingredient of the drug, dosage and frequency should be indicated.
Number of participants taking medication | Throughout study completion, an average of 12 weeks
  During the study, both the increase or reduction of chronic analgesic medication taken by the participant for pain management and the intake of new rescue medication, which is medication taken occasionally for symptomatic or symptom management, treatment of crises or exacerbations, will be recorded.
Knee range of motion (ROM) | Throughout study completion, an average of 12 weeks
  To assess ROM, the participant will be placed in a prone position on a stretcher. An electrogoniometer will then be placed on the leg to be assessed (affected leg) and the participant will be asked to voluntarily flex as far as possible or until pain is felt.
WOMAC scale to measure pain, functional capacity and impact on quality of life | Throughout study completion, an average of 12 weeks
  The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) questionnaire is used to assess participants' perceived clinical changes in knee pain, stiffness and function.
Quality of Life Questionnaire SF-36 | Throughout study completion, an average of 12 weeks
  The SF-36 health questionnaire is composed of 36 items that aim to collect all relevant aspects to characterize the health of an individual.
KOOS Questionnaire for Knee Assessment | Throughout study completion, an average of 12 weeks
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) has been developed as an instrument to assess the patient's opinion of their knee and associated problems. The scores for each dimension are calculated by summing the responses to the relevant questions. The resulting scores are transformed into a scale from 0 to 100.
Sleep quality using the Pittsburgh test | Throughout study completion, an average of 12 weeks
  Sleep quality is assessed using the Pittsburgh sleep quality questionnaire. This questionnaire has 19 self-assessment questions and 5 questions addressed to the roommate or bed partner, with only the first 19 being used to obtain the overall score.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Martínez Noguera, PhD, Study Chair — Research Center for High Performance Sport. Catholic University of Murcia
Locations (1):
- Research Center for High Performance Sport. Catholic University of Murcia, La Ñora, Murcia, Spain

REFERENCES:
- See also: Website — https://investigacion.ucam.edu/vicerrectorado/ciard